CLINICAL TRIAL: NCT01686815
Title: Cross-sectional Study to Compare Glucose and Lipid Metabolism in SMI Subjects Treated With Either Fanapt (Iloperidone), Zyprexa (Olanzapine), or Risperdal (Risperidone)
Brief Title: Cross-Sectional Iloperidone IVGTT
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Maurizio Fava, MD, Vice Chair, Psychiatry, Massachusetts General Hospital
Other Study IDs: CILO522DUSXXT
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Schizophrenia; Serious Mental Illness; Metabolic Syndrome; Insulin Resistance; Glucose Metabolism
Keywords: metabolic side effects; atypical antipsychotics; FSIVGTT
MeSH Terms: conditions — Schizophrenia; Metabolic Syndrome; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Samples will be retained to test IL-6 and other inflammatory markers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Olanzapine: Olanzapine-treated patients with serious mental illness, such as schizophrenia, schizoaffective disorder, bipolar disorder, major depressive disorder, psychosis NOS, delusional disorder or paranoid disorder.
- Risperidone: Risperidone-treated patients with serious mental illness, such as schizophrenia, schizoaffective disorder, bipolar disorder, major depressive disorder, psychosis NOS, delusional disorder or paranoid disorder.
- Iloperidone: Iloperidone-treated patients with serious mental illness, such as schizophrenia, schizoaffective disorder, bipolar disorder, major depressive disorder, psychosis NOS, delusional disorder or paranoid disorder.

SUMMARY:
This study aims to utilize state of the art procedures such as the frequently sampled intravenous glucose tolerance test (FSIVGTT), Bergman's Minimal Model Analysis, lipoprotein analysis, and DEXA scans to demonstrate that a newer agent, iloperidone, is devoid of the metabolic abnormalities associated with other atypical antipsychotic treatments, namely olanzapine and risperidone, and offers an advantage over these other agents.

DETAILED DESCRIPTION:
This one-month research study examines how Fanapt® (iloperidone), Zyprexa® (olanzapine), or Risperdal® (risperidone) affect glucose metabolism in patients with schizophrenia, schizoaffective disorder, bipolar disorder, major depressive disorder, psychosis NOS, delusional disorder or paranoid disorder. This study requires 3 research visits and includes a physical exam, medical history, vitals, an EKG, cognitive testing, psychological rating scales, a DEXA scan, a nutritional assessment, a 3-hour intravenous glucose tolerance test (IVGTT) and a fasting blood draw.

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female ages 18-65 years
2. Capacity to provide informed consent
3. BMI between 20 and 30 kg/m²
4. Diagnosis of a serious mental illness, including schizophrenia, any subtype; schizoaffective disorder, any subtype; major depressive disorder, bipolar disorder, psychosis NOS, delusional disorder and paranoid disorder
5. Treatment with iloperidone, risperidone, or olanzapine for at least 6 months
6. Stable dose of antipsychotic agent for at least one month
7. Well established compliance with out-patient medications and clinically stable
8. Female subjects will be eligible to participate in the study if they are of non-childbearing potential or of child-bearing potential and willing to practice appropriate birth control methods (complete abstinence from sexual intercourse, female sterilization, sterilization of male partner, implants of levonorgestrel, injectable progestogen, oral contraceptives, intrauterine devices, or double barrier methods of contraception using spermicide with either a condom or diaphragm) during the study.

Exclusion Criteria:

1. Inability to provide informed consent
2. Current substance abuse
3. Psychiatrically unstable and/or hospitalized in the past month
4. History of significant and untreated medical illness including severe cardiovascular, hepatic, renal, or untreated thyroid disease; hepatitis; or HIV
5. Current insulin treatment for diabetes
6. Currently taking the following medications: birth control pills containing norgestrol, steroids, thiazide diuretics, or treatment with agents that induce weight loss
7. Intentions of donating blood during or within 30 days of completion of the study.
8. Use of valproate or carbamazepine within four weeks of the study
9. History of immunosuppression
10. Current or recent radiation or chemotherapy treatment for cancer
11. Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will include 60 outpatients between the ages of 18-65 with schizophrenia, schizoaffective disorder, bipolar disorder, major depressive disorder, psychosis NOS, delusional disorder or paranoid disorder. 60 subjects will be screened and 45 will enter the cross-sectional study (15 olanzapine, 15 iloperidone, 15 risperidone-treated subjects matched for BMI).
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2012-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Difference between cohorts in glucose metabolism | Baseline
  Difference between olanzapine- or risperidone-treated subjects, and Iloperidone-treated subjects on glucose metabolism as measured by the FSIVGTT procedure at one time point (Baseline).
Difference between cohorts in triglycerides | Baseline
  Difference between olanzapine- or risperidone-subjects and subjects treated with iloperidone in triglyceride levels measured at one time point (Baseline).
Difference between cohorts on LDL cholesterol | Baseline
  Difference between olanzapine- or risperidone-subjects and subjects treated with iloperidone in LDL cholesterol levels measured at one time point (Baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Fava, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States